CLINICAL TRIAL: NCT03914417
Title: An Investigator-initiated Study to Evaluate Genomic Markers of Immune Infiltration Before and After Treatment of Actinic Keratosis With Imiquimod 3.75% Cream
Brief Title: Genomic Markers Before and After Treatment of Actinic Keratosis With Imiquimod 3.75% Cream
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Principal Investigator, Sharon Rose, Resident, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-1215
Record Dates: First submitted 2017-05-03; First posted 2019-04-16 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Intervention Model Description: Application of imiquimod 3.75% cream to treat actinic keratosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imiquimod 3.75% cream (Experimental): applied topically
  Interventions: Drug: Imiquimod 3.75% Cream

INTERVENTIONS:
Drug: Imiquimod 3.75% Cream — Approximately two weeks after Day 0, the entire treatment area was treated with imiquimod 3.75% cream. Subjects utilized the 2 weeks on, 2 weeks off, 2 weeks on regimen. Subjects were followed every 2 weeks during treatment (week 2, 4 and 6) and then at 4 and 8 weeks post last-imiquimod application (week 10 and 14).

SUMMARY:
The study team had plans to treat approximately 30 subjects. Each subject that had qualified had at least 4-8 visible AKs on the face and/or scalp. At Day 0, one Actinic Keratosis (AK) in the treatment area had been biopsied via a 3 mm punch. The tissue collected was sent to pathology for confirmatory diagnosis as well as genomic analysis. The remaining AKs had been identified, photographed, and documented on a transparency. One of the remaining AKs was designated as the target lesion. The patient returned to the clinic in 7 days (+/- 3) for suture removal. Approximately two weeks after Day 0, the entire treatment area was treated with imiquimod 3.75% cream. Subjects utilized the 2 weeks on, 2 weeks off, 2 weeks on regimen. Subjects were followed every 2 weeks during treatment (week 2, 4 and 6) and then at 4 and 8 weeks post last-imiquimod application (week 10 and 14). At week 14, a biopsy via a 3 mm punch was done of the target lesion. Yet, if the target lesion was no longer present, a biopsy was done at the site where the lesion was previously located.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years old.
* Subjects must be in good general health as confirmed by the medical history.
* Subjects must be able to read, sign, and understand the informed consent.
* Prior to imiquimod therapy, subjects must have at least 4-8 actinic keratoses on the face and/or scalp.
* Subject must be willing to forego any other treatments on the face and/or scalp, including tanning bed use and excessive sun exposure while in the study.
* Subject is willing and able to participate in the study as an outpatient, making frequent visits to the study center during the treatment and follow-up periods and to comply with all study requirements including concomitant medication and other treatment restrictions.
* If subject is a female of childbearing potential she must have a negative urine pregnancy test result prior to study treatment initiation and must agree to use an approved method of birth control while enrolled in the study.

Exclusion Criteria:

* Subjects with a history of melanoma anywhere on the body.
* Subjects with an unstable medical condition as deemed by the clinical investigator.
* Subjects with non-melanoma skin cancer on the face and/or or scalp.
* Subjects with any dermatologic disease in the treatment area that may be exacerbated by the treatment proposed or that might impair the evaluation of AKs.
* Subjects who have previously been treated with imiquimod: on the face or scalp in the past 6 months; or outside of the study area within the past 30 days.
* Women who are pregnant, lactating, or planning to become pregnant during the study period.
* Subjects who have experienced a clinically important medical event within 90 days of the visit (e.g., stroke, myocardial infarction, etc).
* Subjects who have active chemical dependency or alcoholism as assessed by the investigator.
* Subjects who have known allergies to any excipient in the study cream.
* Subjects who are currently participating in another clinical study or have completed another clinical study with an investigational drug or device on the study area within 30 days prior to study treatment initiation.
* Subjects who have received any of the following within 90 days prior to study treatment initiation:

  * interferon or interferon inducers
  * cytotoxic drugs
  * immunomodulators or immunosuppressive therapies (inhaled/ intranasal steroids are permitted)
  * oral or parenteral corticosteroids
  * topical corticosteroids if greater than 2 mg/day
  * any dermatologic procedures or surgeries on the study area (including any AK treatments)
* Subjects who have used any topical prescription medications on the study area within 30 days prior to study treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Rose, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment/Enrollment from Jan 1, 2013 - Jan 1, 2015
Groups:
- Imiquimod 3.75% Cream: Imiquimod 3.75% Cream topically: Approximately two weeks after Day 0, the entire treatment area was treated with imiquimod 3.75% cream. Subjects utilized the 2 weeks on, 2 weeks off, 2 weeks on regimen.
Period: Overall Study
Arm/Group | Imiquimod 3.75% Cream
Started | 21
Completed | 19
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Imiquimod 3.75% Cream
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 73 [65 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders
Description: The number of participants with reduction in number of AKs on the face and/or scalp after application of imiquimod 3.75%.
Time Frame: Day 70
Measure: Count of Participants; unit: Participants
Arm/Group | Imiquimod 3.75% Cream
Number analyzed (Participants) | 19
Participants | 19

2. Secondary Outcome: Number of Treatment Related Adverse Events
Description: The safety of imiquimod 3.75% on the face and/or scalp was determined by the number of treatment related adverse events that occur during the study.
Time Frame: Day 70
Measure: Number; unit: events
Arm/Group | Imiquimod 3.75% Cream
Number analyzed (Participants) | 19
events | 8

ADVERSE EVENTS:
Time Frame: 70 days
Arm/Group | Imiquimod 3.75% Cream
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 16/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imiquimod 3.75% Cream (N=19)
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Left Post-auricular lymphadenopathy (Blood and lymphatic system disorders) | 2
Maculopapular Rash, forearms (Skin and subcutaneous tissue disorders) | 1
Pruritus on treatment area (Skin and subcutaneous tissue disorders) | 2
Arthralgias (Musculoskeletal and connective tissue disorders) | 1
Intolerable LSR (Skin and subcutaneous tissue disorders) | 1
Flu-like symptoms (General disorders) | 2
Viral Upper Respiratory Infection (Infections and infestations) | 2
Facial Swelling (Skin and subcutaneous tissue disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Oral Aphthous Ulcer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fracture of toe (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes